CLINICAL TRIAL: NCT05311748
Title: Prospective Cross-sectional Evaluation of Penile Helicine Circulation by Power Doppler During Dynamic Ultrasound in Veno-occlusive Erectile Dysfunction
Brief Title: Prospective Cross-sectional Evaluation of Penile Helicine Circulation in Veno-occlusive Erectile Dysfunction
Acronym: PD and VOD
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonio Luigi Pastore, PROF, MD, PhD, University of Roma La Sapienza
Other Study IDs: UrolUNIVPISA
Record Dates: First submitted 2022-03-15; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Erectile Dysfunction Due to Arterial Disease
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound and doppler — Penile echocolour doppler ultrasound

SUMMARY:
Background: The aim of this study is to evaluate the usefulness of Power Doppler in order to improve the diagnostic work up of veno-occlusive erectile dysfunction patients.

Materials and Methods: Two hundred and two patients affected by erectile dysfunction, mean IIEF 5 = 13.5 (12-17) for at least 6 months, were enrolled in a prospective cross-sectional study. All patients underwent Dynamic Power Doppler after intracevernous injection of vasoactive drugs. Poor responders patients subsequently underwent to cavernosometry to get a full assessment of the vascular framework.

DETAILED DESCRIPTION:
Veno-occlusive continence is linked both to the integrity of neurological, vascular, and endocrine structures and to the fibro-elastic characteristics of the cavernous tissue. In most subjects with Erectile Dysfunction (ED), the erectile tissue presents histological alterations such as the reduction of smooth muscle cells and the increased deposition of connective tissue. A hypothesis describes these changes as promotors for the onset of veno-occlusive dysfunction (VOD).

Dynamic cavernosometry, supplemented by contrast cavernosography, still represents the gold standard for the diagnosis of VOD allowing the visualization of the competent venous districts. These investigations, which had moderate popularity in the 1980s and underwent several variations in the methodology of execution, are rarely used today due to their invasiveness, the need for dedicated instruments and the scarce success of commonly adopted surgical treatments (vein ligation surgery).

The recent introduction of endovascular techniques sheds new light on the correct classification of vascular ED, especially in those patients with a sub-optimal response to the use of drug therapy as an alternative to prosthetic surgery.

Advances in imaging techniques, including Power Doppler (PD) ultrasonography, allow an accurate and complete study of penile circulation including the study of low-flow vessels.

The introduction of PD, during the penile duplex ultrasound routinely performed, had additionally permitted the extension of the field of the study into the arteriolar circulation of the corpora cavernosa, making possible the assessment of the vessels with a "low speed flow", like the helicine arteries, which escape the standard Doppler Pulsated evaluation; especially during the phases of the penile tumescence and partial rigidity, phases 1-2, according to Erection Hardness Score .

From an anatomical and vascular point of view, the helicine arteries usually describe an acute angle with the cavernous artery, delineating a Cavernous Terminal Unit (CTU).

The dynamic penile echo-color-doppler ultrasound can evaluate the correct assessment of the CTU, by applying the PD function. In fact, the PD module, with calibration of the pulse repetition frequency (PRF) of the transducer at 700 HZ applied to the cavernous arteries in the dynamic phase, allows the study of the ramifications of the arteries up to the 3rd order and their inclination in relation to the main trunk, expression or not of the integrity of the CTU. In this contest, PD applied to dynamic penile duplex ultrasound, has established itself as a method potentially suitable in the assessment of patients with VOD.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients affected by erectile dysfunction for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Echocolour doppler Evaluation of the Index of Maintenance of Erection (n.v. <0.25). | 90 days
  Every subject will be studied by penile ultrasound with color doppler

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Urology Unit, Sapienza University of Rome, Latina
  - Alessandro Zucchi, Pisa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim N, Azadzoi KM, Goldstein I, Saenz de Tejada I. A nitric oxide-like factor mediates nonadrenergic-noncholinergic neurogenic relaxation of penile corpus cavernosum smooth muscle. J Clin Invest. 1991 Jul;88(1):112-8. doi: 10.1172/JCI115266. PMID 1647413